CLINICAL TRIAL: NCT02471820
Title: Phase II Open Label Study for the Assessment of the Efficacy and Safety of Lenalidomide & Adriamycin & Low Dose Dexamethasone (RAD) in Newly Diagnosed, Symptomatic Multiple Myeloma Patients
Brief Title: Lenalidomide & Adriamycin & Dexamethasone (RAD) in Newly Diagnosed, Multiple Myeloma Patients
Acronym: RAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meletios A. Dimopoulos (Other)
Responsible Party: Sponsor-Investigator, Meletios A. Dimopoulos, Professor of Department of Clinical Therapeutics University of Athens School of Medicine, University of Athens
Organization: University of Athens (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-GMSG-392; 2011-001499-20 (EudraCT Number)
Record Dates: First submitted 2015-06-05; First posted 2015-06-15 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Doxorubicin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide, adriamycin & dexamethasone (Experimental): Lenalidomide 25 mg administered orally for the first 21 days of each 28-day-cycle, plus Adriamycin i.v. on days 1,2,3 & 4 of every cycle, plus Dexamethasone 40 mg orally on days 1, 8, 15 & 22 of every cycle for 4 cycles
  Interventions: Drug: Lenalidomide; Drug: Adriamycin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide 25 mg by mouth for the first 21 days of a 28-day-cycle for 4 cycles
  Other Names: Combination of Lenalidomide, adriamycin & dexamethasone
Drug: Adriamycin — Adriamycin as intravenous bolus infusion at a dose of 9 mg/m2, on days 1-4 of a 28-day cycle for 4 cycles
  Other Names: Combination of Lenalidomide, adriamycin & dexamethasone
Drug: Dexamethasone — Dexamethasone by mouth at a dose of 40 mg, on days 1, 8, 15, and 22 of a 28-day cycle for 4 cycles
  Other Names: Combination of Lenalidomide, adriamycin & dexamethasone

SUMMARY:
This study is to assess the efficacy and safety of lenalidomide in combination with adriamycin and low dose dexamethasone in newly diagnosed patients with symptomatic multiple myeloma as well as to collect information regarding the effect of this regimen on angiogenesis and bone remodeling of the study population.

DETAILED DESCRIPTION:
This is a Phase II, non randomized, non- comparative, open label trial which assess the efficacy and safety of lenalidomide, adriamycin and low dose dexamethasone combination (RAD) in 45 newly diagnosed patients with symptomatic multiple myeloma as well as to collect information regarding the effect of this regimen on angiogenesis and bone remodeling of the study population. The recruitment period is estimated for 5 months while the treatment period and the follow up period 4 months and 1 month respectively. During the treatment initiation visit the response to the combination RAD according the International Myeloma Working Group (IMWG) criteria will be evaluated, biochemical markers of bone metabolism and angiogenic cytokines will be measured as well. IMWG Response evaluation will be repeated the day 1 of each treatment cycle as well as at the response evaluation visit. Finally biochemical markers of bone metabolism and angiogenic cytokines will be measured once more at the end of treatment visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to read and understand the Informed Consent Form (ICF).
2. Subjects willing to participate in the study and comply with its procedures.
3. Subjects who have signed the ICF
4. Newly diagnosed patients with symptomatic MM according to the criteria of IMWG
5. Subjects eligible for autologous stem cell transplantation
6. Age 18-70 years, of either sex
7. karnofsky ≥ 60
8. Platelets ≥ 100x109/L
9. Neutrophils ≥ 1.5x109/L
10. Alanine transaminase (ALT) & Aspartate transaminase (AST) ≤ 3-fold of upper normal limit
11. Bilirubin ≤ 2-fold of upper normal limit
12. Creatinine clearance ≥60 ml/min
13. Expected survival ≥ 6 months as per PI's clinical judgment
14. Subjects able to tolerate aspirin, low molecular weight heparin or coumarinic agents as prophylactic anticoagulation
15. Female subject of childbearing potential must have 2 negative serum pregnancy tests (hCG) at Screening (once within 10-14 days and once 24 h before the study drug administration) and if sexually active must be using two medically acceptable, highly effective, adequate forms of birth control (ie, failure rate <1% per year when used consistently and correctly) prior to Screening and and for time period at least 28 days before the study drug administration and agree to continue using it while being in the study (Screening and Treatment Periods including dose interruptions). A female subject should continue using a highly effective method of birth control for 30 days following the end of treatment.
16. A male subject must agree to use an adequate form of contraception for the duration of the study, while taking the study drug, during dose interruptions at for at least 28 days after the last dose of study drug even if he has had a successful vasectomy and agree to have sexual relations only with women who use a highly effective birth control method.
17. Subjects must be free of any clinically significant disease (other than MM) that would interfere with study evaluations

Exclusion Criteria:

1. Pregnancy, breastfeeding οr intention of pregnancy during the trial
2. Suspected or known hypersensitivity to any of the study drugs
3. Ongoing severe infection requiring intravenous antibiotic treatment
4. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer from which the subject has been disease-free for at least 5 years. Concurrent prostate cancer for which the patient is receiving therapy will not be considered an exclusion if the Prostatic specific antigen (PSA) has been stable for 3 years
5. Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia
6. Myocardial infraction within 6 months before enrollment, New York Heart Association (NYHA) Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmia, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
7. Uncontrolled medical problems such as diabetes, coronary artery disease, hypertension, unstable angina, arrhythmia, pulmonary, hepatic and renal diseases unless renal insufficiency is considered to be secondary to MM
8. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the ICF
9. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she will participate in the study or confounds the ability to interpret data from the study
10. Subjects with any clinical condition that would affect study's outcome
11. Participation in another interventional clinical trial in the 4 weeks preceding enrollment or planning to participate in another interventional clinical trial during the planned period of this study, except of the clinical trials that implicate drugs of supportive treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 142 days
  Assessment of the overall response rate of study population to RAD regimen (including stringent complete response, complete response, very good partial response, partial response and stable disease) according to the uniform criteria of IMWG (International Myeloma Working Group) regarding the response to multiple myeloma therapy

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 142 days
Time to progression (TTP) | 142 days
Time to Next Therapy (TtNT) | 142 days
Number and severity of Adverse events as a measure of safety and toxicity profile | 142 days
  Adverse events will be assessed at each visit and graded according to the National Cancer Institute Common Toxicity Criteria (version 2.0)

OTHER OUTCOMES:
Number of stem cell collected before Autologous Stem Cell Transplantation (ASCT) | 142 days
Dickkopf-1 (DKK-1) | 1 day
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Dickkopf-1 (DKK-1) | 112 days
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
C-telopeptide of type-I collagen (CTX) | 1 day
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
C-telopeptide of type-I collagen (CTX) | 112 days
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Tartrate-resistant acid phosphatase isoform-5b (TRACP-5b) | 1 days
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Tartrate-resistant acid phosphatase isoform-5b (TRACP-5b) | 112 days
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Bone-alkaline phosphatase (bALP) | 1 day
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Bone-alkaline phosphatase (bALP) | 112 days
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Osteocalcin (OC) | 1 day
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Osteocalcin (OC) | 112 days
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
C-terminal propeptide of procollagen type-I (CICP) | 1 day
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
C-terminal propeptide of procollagen type-I (CICP) | 112 days
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Soluble and total RANKL (sRANKL, tRANKL) | 1 day
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Soluble and total RANKL (sRANKL, tRANKL) | 112 days
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Osteoprotegerin (OPG) | 1 day
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Osteoprotegerin (OPG) | 112 days
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Osteopontin (OPN) | 1 day
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Osteopontin (OPN) | 112 days
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Macrophage inflammatory protein 1-alpha (MIP-1α) | 1 day
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Macrophage inflammatory protein 1-alpha (MIP-1α) | 112 days
  Biochemical markers of bone remodeling will be measured in the serum of patients at therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Angiopoietin-1 & -2 | 1 day
  Angiogenic cytokines, which will be evaluated in the serum of patients during therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Angiopoietin-1 & -2 | 112 days
  Angiogenic cytokines, which will be evaluated in the serum of patients during therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Angiogenin | 1 day
  Angiogenic cytokines, which will be evaluated in the serum of patients during therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Angiogenin | 112 days
  Angiogenic cytokines, which will be evaluated in the serum of patients during therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
VEGF | 1 day
  Angiogenic cytokines, which will be evaluated in the serum of patients during therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
Vascular endothelial growth factor (VEGF) | 112 days
  Angiogenic cytokines, which will be evaluated in the serum of patients during therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
VEGF-A | 1 day
  Angiogenic cytokines, which will be evaluated in the serum of patients during therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
VEGF-A | 112 days
  Angiogenic cytokines, which will be evaluated in the serum of patients during therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
basic fibroblast growth factor (bFGF) | 1 day
  Angiogenic cytokines, which will be evaluated in the serum of patients during therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle
basic fibroblast growth factor (bFGF) | 112 days
  Angiogenic cytokines, which will be evaluated in the serum of patients during therapy commencement on Day 1 of cycle 1 and at therapy completion on day 28 of cycle 4. 28-days-cycle

CONTACTS AND LOCATIONS:
Overall Officials: Meletios Dimopoulos, Doctor, Principal Investigator — General Hospital of Athens "Alexandra"; Eirini Katodritou, Doctor, Principal Investigator — Theageneio Anticancer Hospital of Thessaloniki; Nikolaos Anagnostopoulos, Doctor, Principal Investigator — General Hospital of Athens "G. Gennimatas''; Argirios Symeonidis, Doctor, Principal Investigator — University General Hospital of Patras
Locations (4):
- Greece (4):
  - General Hospital of Athens "G. Gennimatas", Athens, Attica
  - General Hospital of Athens "Alexandra", Athens, Attica
  - University General Hospital of Patras, Pátrai, Patra
  - Theageneio Anticancer Hospital of Thessaloniki, Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided